CLINICAL TRIAL: NCT00301119
Title: NYU Lung Cancer Biomarker Center
Brief Title: Lung Cancer Biomarkers and Screening
Acronym: NYULCBC
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 8896; NYU-H-8896-06-B; NCT00212524 (obsolete NCT alias)
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: small cell lung cancer; non-small cell lung cancer; smoker lung cancer screening; low dose spiral CT screening
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood serum, plasma, urine, sputum, BAL, lung tissue, buccal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lung cancer screening cohort: observational only. no intervention. current, former and never smokers over age 50 without history of cancer, except for non melanoma skin cancer, no previous treatment with chemotherapy.
- r/o lung cancer: observational only. no intervention. patients with CT findings suspicious for lung cancer who are undergoing bronchoscopy and/or surgery.

SUMMARY:
RATIONALE: Screening tests that use biomarkers may help doctors find tumor cells early and plan effective treatment for lung cancer.

PURPOSE: This clinical trial is studying biomarkers in screening participants for lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify and validate biomarkers for the early detection of lung cancer in individuals at low- or high-risk for smoking-related cancers.
* Identify preneoplastic cellular changes and lesions in these patients.

OUTLINE: Participants are stratified according to lung cancer risk status (with or without increased risk).

Group 1 (screening cohort): Participants complete a questionnaire and undergo pulmonary function testing, multidetector chest CT scan, sputum induction, and phlebotomy.

Group 2 (rule-out lung cancer): Participants complete the same questionnaire and undergo the same tests and scans as in group 1. Some participants may undergo fiberoptic bronchoscopy based upon CT scan results with transbronchial or endobronchial biopsies. Some participants may undergo lung resection. Tissue samples are collected from surgery or biopsy.

PROJECTED ACCRUAL: A total of participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Screening Cohort

  * At high- or low-risk for lung cancer
  * Smoking history ≥ 20 pack years*

    * With or without workplace exposure to asbestos
* NOTE: * Participants with < 20 pack years of smoking are eligible if 50 years of age or older
* Rule-Out Lung cancer group

  * Referred for evaluation of suspicious nodules with 1 of the following diagnoses:

    * Lung cancer
    * Nonmalignant nodules (control group)

PATIENT CHARACTERISTICS:

* Not pregnant
* No prior malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects at risk for lung cancer and controls from community, private physician referrals, local trade unions, employee health fairs, word of mouth and print advertisements.
  patient referrals from physician outpatient offices and inpatients with CT findings suspicious for lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10850 (Estimated)
Dates: Start 2000-05; Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Lung cancer diagnosis as measured by CT scan findings and pathology findings annually | 07/01/2015

SECONDARY OUTCOMES:
Precancerous lung nodules as measured by CT scan findings and pathology findings annually | 07/01/2015

CONTACTS AND LOCATIONS:
Overall Officials: James J. Tsay, MD, MSc, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cancer Institute at New York University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Greenberg AK, Rimal B, Felner K, Zafar S, Hung J, Eylers E, Phalan B, Zhang M, Goldberg JD, Crawford B, Rom WN, Naidich D, Merali S. S-adenosylmethionine as a biomarker for the early detection of lung cancer. Chest. 2007 Oct;132(4):1247-52. doi: 10.1378/chest.07-0622. PMID 17934114
- [Result] Greenberg AK, Lu F, Goldberg JD, Eylers E, Tsay JC, Yie TA, Naidich D, McGuinness G, Pass H, Tchou-Wong KM, Addrizzo-Harris D, Chachoua A, Crawford B, Rom WN. CT scan screening for lung cancer: risk factors for nodules and malignancy in a high-risk urban cohort. PLoS One. 2012;7(7):e39403. doi: 10.1371/journal.pone.0039403. Epub 2012 Jul 2. PMID 22768300
- [Result] Rom WN, Goldberg JD, Addrizzo-Harris D, Watson HN, Khilkin M, Greenberg AK, Naidich DP, Crawford B, Eylers E, Liu D, Tan EM. Identification of an autoantibody panel to separate lung cancer from smokers and nonsmokers. BMC Cancer. 2010 May 26;10:234. doi: 10.1186/1471-2407-10-234. PMID 20504322